CLINICAL TRIAL: NCT04705064
Title: Development and Prospective Validation of an Artificial Intelligence Model to Predict Postoperative Acute Kidney Injury
Brief Title: Artificial Intelligence and Postoperative Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyung-Chul Lee, Assistant professor, Seoul National University Hospital
Other Study IDs: 2012-069-1180
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Non-cardiac Surgery
Keywords: Artificial Intelligence; Postoperative acute kidney injury; Prospective validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AI_AKI: Adults patients undergoing non-cardiac surgery
  Interventions: Diagnostic Test: Prediction of postoperative acute kidney injury using an artificial intelligence

INTERVENTIONS:
Diagnostic Test: Prediction of postoperative acute kidney injury using an artificial intelligence — The performance of an artificial intelligence model to predict postoperative acute kidney injury will be tested prospectively.

SUMMARY:
The main objective of this study is to develop and validate an artificial intelligence model that predicts postoperative acute kidney injury.

DETAILED DESCRIPTION:
Postoperative acute kidney injury is known to increase the length of hospital stay and healthcare cost. A lot of risk prediction models have been developed for identifying patients at increased risk of postoperative acute kidney injury. Recent advances in artificial intelligence make it possible to manage and analyze big data. Prediction model using an artificial intelligence and large-scale data can improve the accuracy of prediction performance. Furthermore, the use of an artificial intelligence may be a useful adjuvant tool in making clinical decisions or real-time prediction if it is integrated into the electrical medical record systems. However, before implementing an artificial intelligence model into the clinical setting, prospective evaluation of an artificial intelligence model's real performance is essential. However, to our knowledge, there was no artificial intelligence model for prediction of postoperative acute kidney injury, which was prospectively evaluated. Therefore, we aimed to develop an artificial intelligence model which predicts postoperative acute kidney injury and evaluate the model's performance prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients undergoing non-cardiac surgery

Exclusion Criteria:

* Age under 18 years
* Surgery duration < 1 hour
* Transplantation surgery
* Nephrectomy
* Cardiac surgery
* Patients who had severe kidney dysfunction preoperatively as follows:
* Serum creatinine ≥ 4 mg/dl
* Estimated glomerular filtration rate <15 ml/min/1.73m2
* History of renal replacement therapy
* Patients who had no results of preoperative or postoperative serum creatinine

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults patients undergoing non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of postoperative acute kidney injury | during the postoperative seven days
  postoperative acute kidney injury (diagnosed by KDIGO criteria using peak serum creatinine level) included all acute kidney injury events regardless of acute kidney injury severity

CONTACTS AND LOCATIONS:
Locations (1):
- Hyung-Chul Lee, Seoul, South Korea